CLINICAL TRIAL: NCT04542603
Title: Neuroinflammation and Age-associated Brain Pathology: Two Potential Mechanisms of Cognitive Impairment in Ovarian Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No recruitment/enrollment and funding expired.
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Jonathan E McConathy, M.D. P.h.D., Director for the Division Molecular Imaging and Therapeutics Affiliation: University of Alabama at Birmingham Collaborators:, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: R20-100
Record Dates: First submitted 2020-08-13; First posted 2020-09-09 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — 2-(4'-(methylamino)phenyl)-6-hydroxybenzothiazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- treatment naivete women with stage 1-4 newly diagnosed ovarian (Experimental)
  Interventions: Drug: [11C]PiB and 18F-labeled DPA-714 PET scan

INTERVENTIONS:
Drug: [11C]PiB and 18F-labeled DPA-714 PET scan — One PET with [11C]PiB and One PET with [18F]DPA-714 before chemotherapy treatment begins. One more PET with [18F]DPA-714 after completion of 3-6 cycles of chemotherapy.

SUMMARY:
This clinical study will use the small molecule translocator protein (TSPO) ligand, 18F-labeled DPA- 714, to visualize and quantify neuroinflammation in treatment naivete women with stage 1-4 newly diagnosed ovarian cancer (without brain metastases) prior to starting neoadjuvant chemotherapy treatment (baseline) and within a month of completing first 6 cycles of cytotoxic chemotherapy treatment (follow-up). In addition, we will use the well-characterized small molecule PET(Positron Emission Tomography) tracer, 11C-labeled Pittsburgh compound B (PiB) to visualize and quantify the regional brain distribution of pathological amyloid deposition at baseline only. The brain amyloid PET and MRI data acquired through this study will be correlated with cognitive test data, clinical data, genetic testing, and biospecimens collected in this study.

ELIGIBILITY:
Inclusion Criteria:

1. 50 years of age or older
2. Female gender
3. Newly diagnosed treatment naïve women with stage III/IV epithelial ovarian cancer (without known brain metastases).
4. High or mixed affinity binder for TSPO ligands based on genotyping for single nucleotide polymorphism (SNP) rs6971.
5. English is primary language
6. Planned neoadjuvant chemotherapy with platinum and taxane drugs

Exclusion Criteria:

1. Contraindication to MRI
2. Pregnancy
3. Lactation
4. Individuals who are unable to participate in the imaging portion due to severity of their medical condition
5. Chronic infectious disease (e.g. HIV, HCV)
6. Chronic inflammatory disease (e.g., fibromyalgia, MS, etc) or autoimmune disease
7. Viral or bacterial illness requiring medical attention and/or antibiotics within 1 month of study participation
8. Blood or blood clotting disorder
9. Cancer that has metastasized to the brain
10. Positive urine hCG test day of procedure or a serum hCG test within 48 hours prior to the administration of [18F]DPA-714 and [11C]PiB.
11. Currently enrolled in a clinical trial utilizing experimental therapies.
12. Low affinity binder for TSPO ligands based on genotyping for SNP rs6971.
13. Prior brain tumor or other neurological condition known to affect cognition
14. A diagnosis of dementia unrelated to cancer or an adjusted MMSE score < 24

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-06 (Estimated); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Measure neuroinflammation by calculating the concentration and regional distribution of activated brain microglia/macrophages using the PET ligand [F-18]DPA-714. | Pre-study visit through 3-6 cycles of chemotherapy (each cycle is typically 2 weeks)

SECONDARY OUTCOMES:
Correlate cognitive impairment before and after beginning cancer therapy with the concentration and regional brain distribution of pathologic amyloid deposition measured with the PET tracer [C-11]PiB prior to beginning therapy. | Pre-study visit through 3-6 cycles of chemotherapy (each cycle is typically 2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan McConathy, MD, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: No
To be determined